CLINICAL TRIAL: NCT02683798
Title: Comparison of Two Weight Loss Maintenance Interventions in Counterweight Plus
Brief Title: BEYOND Weight Loss Maintenance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN15HN592
Record Dates: First submitted 2016-02-09; First posted 2016-02-17 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Obesity
Keywords: Weight loss maintenance
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous energy restriction (Active Comparator): 1 x formula food (202-209kcal) meal replacement per day
  Interventions: Dietary Supplement: Continuous energy restriction
- Intermittent energy restriction (Experimental): 4 x formula food (202-209kcal) total diet replacement per day, on 2 days per week
  Interventions: Dietary Supplement: Intermittent energy restriction

INTERVENTIONS:
Dietary Supplement: Continuous energy restriction — 1 x formula food (202-209kcal) meal replacement per day
  Arms: Continuous energy restriction
Dietary Supplement: Intermittent energy restriction — 4 x formula food (202-209kcal) total diet replacement per day, on 2 days per week
  Arms: Intermittent energy restriction

SUMMARY:
A study to determine the effectiveness of two weight loss maintenance interventions in Counterweight Plus, a structured weight management programme.

DETAILED DESCRIPTION:
Introduction: Long-term maintenance of non-surgical weight loss remains the most significant problem in obesity treatment. This study will compare the effectiveness of two different weight loss maintenance strategies used as part of the Counterweight Plus weight management programme. This study will also evaluate the behavioural impact of the Counterweight Plus interventions and include process evaluations and cost analysis.

Methods: 80 patients and 10 practitioners will be recruited into the study. Main inclusion criteria for patients are:

Completed Counterweight Plus, which includes 12-20 weeks total diet replacement (TDR), 8 weeks food reintroduction (FR) and achieved >10kg weight loss. All participants will be followed up for 18 months in total.

Results: The primary outcome of this study is the difference in weight change between the two groups at 6 months. Frequency of use of behavioural strategy will be quantified for both practitioners and patients during voice recorded consultations. The relationship between weight change and the use of behavioural strategy will be assessed.

Hypothesis: This study will establish if the novel intermittent use of formula diet strategy is more effective at preventing weight regain in comparison to usual care. It will also provide evidence of the frequency of use of behavioural strategies within routine Counterweight Plus delivery, as well as establishing the cost of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Completed Counterweight Plus Total Diet Replacement and Food Reintroduction stages and achieved >10kg weight loss

Exclusion Criteria:

* People currently participating in another clinical research trial (not including BEYOND Weight Loss study)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Weight change | Baseline, 26 weeks
  Difference between the two groups in change in body weight (kg)

SECONDARY OUTCOMES:
Weight change | Baseline, 52 weeks, 78 weeks
  Change in body weight (kg)
Acceptability | Baseline, 26 weeks, 52 weeks, 78 weeks
  Number of clinic appointments attended as a proportion of the total number offered
Behavioural strategies | 78 weeks
  Number of times behaviour change strategies used, assessed by qualitative analysis/coding of consultations
Eating behaviours | Baseline, 26 weeks, 52 weeks, 78 weeks
  Change measured using Three Factor Eating Questionnaire- R18 (TFEQ-R18)
Quality of life | Baseline, 26 weeks, 52 weeks, 78 weeks
  Change measured using EuroQoL-5D (EQ-5D)
Cost of interventions | 78 weeks
  Difference between groups

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lean, FRCPS, Principal Investigator — University of Glasgow
Locations (3):
- United Kingdom (3):
  - NHS Lothian, Edinburgh
  - NHS Greater Glasgow and Clyde, Glasgow
  - NHS Highland, Inverness

REFERENCES:
- [Derived] Brosnahan N, Hankey C, Leeds A, Leslie W, Thom G, Hutchison L, Govan L, Ross H, Lean MEJ. Diet strategies for maintaining substantial therapeutic weight loss: 78-week mixed methods randomised trial. Clin Nutr. 2025 Oct;53:188-198. doi: 10.1016/j.clnu.2025.08.009. Epub 2025 Aug 12. PMID 40934815